CLINICAL TRIAL: NCT06227052
Title: Vapocoolant Application for Pain Reduction During Office-based Gynecologic Procedures: a Randomized Controlled Trial (VAPOR)
Brief Title: Applying Num Vapocoolant Spray to Cervix Before Paracervical Block to Decrease Pain During Gynecology Procedures
Acronym: VAPOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: Lakshmi Devi and Devraj Sharma Endowment (Unknown)
Responsible Party: Principal Investigator, Catherine Rault, Complex Family Planning Fellow, Queen's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RA-2023-046 VAPOR1004
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pain With Paracervical Block; Pain With Gynecology Procedure; Pain
Keywords: Pain with Paracervical Block; Pain with Gynecology Procedure; Num Vapocoolant Spray; Vapocoolant Spray; Vapocoolant
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Research coordinators who will be collecting pain scales from patients will be blinded to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Natures Tears (Placebo Comparator): This is the placebo arm. Participants in this arm will receive Natures Tears spray during their gynecologic procedure. They will receive the spray on their cervix right before the paracervical block. Natures Tears is normal saline, which is sprayed from a canister similar to the Num vapocoolant.
  Interventions: Other: Placebo
- Num Vapocoolant Spray (Experimental): This is the intervention arm.
  Interventions: Device: Num Vapocoolant Spray

INTERVENTIONS:
Device: Num Vapocoolant Spray — This is the study arm. Partipants in this arm will receive Num vapocoolant spray during their gynecologic procedure. They will receive the spray on their cervix right before the paracervical block. Num Vapocoolant spray is currently FDA approved to be used on skin prior to injections. The investigators are using it in the same fashion but in the vagina on the cervix to help with the pain of the paracervical block injection.
  Arms: Num Vapocoolant Spray
Other: Placebo — This is the placebo. This group will receive Natures tear normal saline spray.
  Arms: Natures Tears

SUMMARY:
The purpose of this study is to assess if Num vapocoolant spray decreases pain associated with paracervical block in gynecology procedures.

DETAILED DESCRIPTION:
After patients seen in our clinic have decided to proceed with a gynecology procedure that requires a paracervical block, the doctor will evaluate if the patient meets eligibility criteria for this study. If the patient does meet eligibility criteria, the doctor will inform the patient about the study and the potential risks. All patients will be given written informed consent. If the patient decides to participate in the study, they will be randomized (patient blinded) to receive either Num vapocoolant spray or placebo (normal saline spray), which the patient will receive during their gynecologic procedure just before the paracervical block. The purpose of this study is to see if the Num vapocoolant spray decreases patients pain with the paracervical block.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older

Undergoing a procedure requiring paracervical block

English-speaking

Able and willing to sign the informed consent form and agree to terms of the study

Exclusion Criteria:

* Required or requested narcotics, anxiolytics, IV sedation, or general anesthesia for the procedure

Declines or has a contraindication/allergy to ibuprofen

Previously received vapocoolant spray in a medical setting

Contraindications or allergies to lidocaine for paracervical block or vapocoolant spray components (1,1,3,3-pentafluoropropaine or 1,1,1,2-tetrafluroethane)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Tschann, PhD, Study Chair — University of Hawaii
Locations (1):
- Queens Medical Center POB1 Clinic 1004, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact corresponding author regarding access to IPD.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: If interested, please contact corresponding author to access IPD.
Access Criteria: Criteria for accessing IPD will be established at the conclusion of the study.
URL: https://www.fprchawaii.org/

REFERENCES:
- [Background] Lambert T, Truong T, Gray B. Pain perception with cervical tenaculum placement during intrauterine device insertion: a randomised controlled trial. BMJ Sex Reprod Health. 2020 Apr;46(2):126-131. doi: 10.1136/bmjsrh-2019-200376. Epub 2019 Oct 30. PMID 31666302
- [Background] Kosaraju A, Vandewalle KS. A comparison of a refrigerant and a topical anesthetic gel as preinjection anesthetics: a clinical evaluation. J Am Dent Assoc. 2009 Jan;140(1):68-72; quiz 112-3. doi: 10.14219/jada.archive.2009.0020. PMID 19119169
- [Background] DiMarco AC, Wetmore AO. Clinical Comparison: Fast-Acting and Traditional Topical Dental Anesthetic. Anesth Prog. 2016 Summer;63(2):55-61. doi: 10.2344/0003-3006-63.2.55. PMID 27269661
- [Background] Zhu Y, Peng X, Wang S, Chen W, Liu C, Guo B, Zhao L, Gao Y, Wang K, Lou F. Vapocoolant spray versus placebo spray/no treatment for reducing pain from intravenous cannulation: A meta-analysis of randomized controlled trials. Am J Emerg Med. 2018 Nov;36(11):2085-2092. doi: 10.1016/j.ajem.2018.03.068. Epub 2018 Mar 27. PMID 30253890
- [Background] Isik MT, Oztunc G. Effects of subcutaneous injection after coolant spray on pain, hematoma, and ecchymosis in three different regions. Nurs Forum. 2022 May;57(3):352-357. doi: 10.1111/nuf.12688. Epub 2021 Dec 30. PMID 34970741
- [Background] Wang L, Fang L, Zhou Y, Fang X, Liu J, Qu G. Efficacy and safety of vapocoolant spray for vascular puncture in children and adults: A systematic review and meta-analysis. PLoS One. 2023 Feb 13;18(2):e0279463. doi: 10.1371/journal.pone.0279463. eCollection 2023. PMID 36780438
- [Background] Selvi F, Bedel C, Akcimen M. Evaluation of vapocoolant spray effect on pain reduction during digital nerve block: A randomized clinical trial. Am J Emerg Med. 2021 Dec;50:260-263. doi: 10.1016/j.ajem.2021.08.001. Epub 2021 Aug 6. PMID 34418716
- [Background] Ganji Z, Shirvani MA, Rezaei-Abhari F, Danesh M. The effect of intermittent local heat and cold on labor pain and child birth outcome. Iran J Nurs Midwifery Res. 2013 Jul;18(4):298-303. PMID 24403926
- [Background] Ernst E, Fialka V. Ice freezes pain? A review of the clinical effectiveness of analgesic cold therapy. J Pain Symptom Manage. 1994 Jan;9(1):56-9. doi: 10.1016/0885-3924(94)90150-3. PMID 8169463
- [Background] Unal N, Tosun B, Aslan O, Tunay S. Effects of Vapocoolant Spray Prior to SC LMWH Injection: An Experimental Study. Clin Nurs Res. 2021 Feb;30(2):127-134. doi: 10.1177/1054773818825486. Epub 2019 Jan 30. PMID 30698458
- [Background] Goldthwaite LM, Baldwin MK, Page J, Micks EA, Nichols MD, Edelman AB, Bednarek PH. Comparison of interventions for pain control with tenaculum placement: a randomized clinical trial. Contraception. 2014 Mar;89(3):229-33. doi: 10.1016/j.contraception.2013.11.018. Epub 2013 Dec 10. PMID 24405796
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman AB. Pain control in first-trimester surgical abortion: a systematic review of randomized controlled trials. Contraception. 2010 May;81(5):372-88. doi: 10.1016/j.contraception.2009.12.008. Epub 2010 Jan 27. PMID 20399943
- [Background] Renner RM, Nichols MD, Jensen JT, Li H, Edelman AB. Paracervical block for pain control in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2012 May;119(5):1030-7. doi: 10.1097/AOG.0b013e318250b13e. PMID 22525915
- [Background] Chin J, Kaneshiro B, Elia J, Raidoo S, Savala M, Soon R. Buffered lidocaine for paracervical blocks in first-trimester abortions: a randomized controlled trial. Contracept X. 2020 Oct 18;2:100044. doi: 10.1016/j.conx.2020.100044. eCollection 2020. PMID 33196038
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Renner RM, Edelman AB, Nichols MD, Jensen JT, Lim JY, Bednarek PH. Refining paracervical block techniques for pain control in first trimester surgical abortion: a randomized controlled noninferiority trial. Contraception. 2016 Nov;94(5):461-466. doi: 10.1016/j.contraception.2016.05.005. Epub 2016 May 25. PMID 27235677
- See also: Num Vapocoolant Website — https://623medical.com/.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natures Tears | Num Vapocoolant Spray
Started | 49 | 49
Completed | 48 | 49
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natures Tears | Num Vapocoolant Spray | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.9 (6.7) | 29.7 (6.1) | 29.3 (6.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gestational age [Mean (Standard Deviation); unit: days] | 62.6 (18.8) | 60.2 (16.6) | 61.4 (17.3)
Parity [Count of Participants; unit: Participants] | 33 | 31 | 64
History of vaginal deliveries (1 or more) [Count of Participants; unit: Participants] | 27 | 27 | 54
History of cesarean section (1 or more) [Count of Participants; unit: Participants] | 8 | 10 | 18
History of moderate or severe menstrual cramps [Count of Participants; unit: Participants] | 15 | 19 | 34
Prior gynecologic procedures [Count of Participants; unit: Participants] | 20 | 29 | 49
Anxiety [Count of Participants; unit: Participants] | 14 | 18 | 32
Depression [Count of Participants; unit: Participants] | 9 | 8 | 17
Level of provider [Count of Participants; unit: Participants]
  Intern | 8 | 10 | 18
  resident | 1 | 5 | 6
  fellow | 29 | 30 | 59
  attending | 11 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pain With Paracervical Block
Description: The investigators will ask patients to rate their pain with the paracervical block using a visual analog scale (VAS). The visual analog scale is 100 mm line, with values 0 to 100. 0 is marked as no pain, 100 is marked as worst pain.
Time Frame: Immediately after paracervical block (0 minutes after PCB completed)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Natures Tears | Num Vapocoolant Spray
Number analyzed (Participants) | 48 | 49
units on a scale | 27 [10 to 49] | 20 [5 to 49]

2. Secondary Outcome: Patient Satisfaction With Procedure
Description: The investigators will also ask patients after their gynecologic procedure how satisfied they were with the procedure and the pain control during the procedure using a Visual Analog Scale (VAS). The visual analog scale is 100 mm line, with values 0 to 100. 0 is marked as not satisfied, 100 is marked as extremely satisfied.
Time Frame: Immediately after their gynecologic procedure (0 minutes after procedure completed)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Natures Tears | Num Vapocoolant Spray
Number analyzed (Participants) | 48 | 49
units on a scale
  Satisfaction w procedure | 91.5 [66 to 99] | 94 [74 to 99]
  Satisfaction with pain control during procedure | 82 [48.8 to 98] | 75 [53 to 98.5]

3. Secondary Outcome: Provider Ease of Use
Description: Immediately after the patients gynecologic procedure, the research coordinators will ask the provider how easy it was to use the spray. The provider will use a visual analog scale. The visual analog scale is 100 mm line, with values 0 to 100. 0 is marked as not easy to use, 100 is marked as easy to use.
Time Frame: Within 5 minutes after patient procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Natures Tears | Num Vapocoolant Spray
Number analyzed (Participants) | 48 | 49
units on a scale | 0 [0 to 2] | 0 [0 to 6]

4. Secondary Outcome: Other Pain Points During Gynecology Procedure
Description: The investigators will also look at a patients reported pain using the Visual Analog Scale (VAS) during other times of the procedure. Specifically: Prior to the start of the procedure (baseline) After tenaculum placement, Five minutes post-procedure. The visual analog scale is 100 mm line, with values 0 to 100. 0 is marked as no pain, 100 is marked as worst pain.
Time Frame: Baseline pain (immediately before procedure), after tenaculum (0 minutes after tenaculum placed), and 5 minutes after procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Natures Tears | Num Vapocoolant Spray
Number analyzed (Participants) | 48 | 49
units on a scale
  Baseline Pain | 1 [0 to 3.75] | 0 [0 to 4]
  Tenaculum | 17 [2 to 33] | 9 [1.5 to 24]
  Pain immediately after procedure | 53 [20 to 73.5] | 56 [27 to 72]
  Pain 5 minutes post op | 23 [5.5 to 46.5] | 23 [5.5 to 46.5]

5. Secondary Outcome: Pre Procedure Anxiety
Description: The investigators will also ask the patient how anxious they are before the procedure using the Visual Analog Scale (VAS). The visual analog scale is 100 mm line, with values 0 to 100. 0 is marked as no anxiety, 100 is marked as anxious.
Time Frame: Immediately after enrollment - before procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Natures Tears | Num Vapocoolant Spray
Number analyzed (Participants) | 48 | 49
units on a scale | 59 [35 to 79.8] | 48 [21 to 57]

ADVERSE EVENTS:
Time Frame: 1 week postprocedure
Description: Adverse events were captured in a few ways:
  1. Patients were called 2 days after procedure to see if they had any concerning side effect/symptoms.
  2. If any patients called post op with any concerning side effects/symptoms. All patients were given our clinic line, our 24 hour line to a doctor on call on our team and the research line.
  3. I any patients presented to the ED for complications from procedure.
Arm/Group | Natures Tears | Num Vapocoolant Spray
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 0/48 | 2/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natures Tears (N=48) | Num Vapocoolant Spray (N=49)
Vaginal itching (Reproductive system and breast disorders) | 0 (0) | 1 (1) — ED with vaginal itching for 2 days, prescribed clotrimazole/betamethasone. CT test positive after ED. Rx sent in by us as part of follow up for AE.
Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) — D&C complicated by hemorrhage and re-aspiration. Pt received misoprostol 800 mcg for bleeding in second procedure. Patient tolerated both procedures. Vital signs stable. Hemostasis noted after both initial procedure and re-aspiration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT06227052/Prot_SAP_002.pdf
  • Informed Consent Form (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT06227052/ICF_003.pdf